CLINICAL TRIAL: NCT07244354
Title: Maternal Hypothermia After Caesarean Section - Implications for Postoperative Recovery
Status: Not yet recruiting | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Elizabeth Reine, Professional development and research nurse, Oslo University Hospital
Other Study IDs: 911621
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Caesarean Section
Keywords: patient reported outcome measures; quality of care; patient satisfaction; perioperative hypothermia; post caesarean infection
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Self report questionnaire — No intervention

SUMMARY:
The aim of the study is to assess patient reported outcomes after caesarean section using self report questionnaire.

DETAILED DESCRIPTION:
The project consists of two studies: Study 1 explores patient reported outcomes after caesarean section related to recovery and quality of care. Study 2 explores possible associations between perioperative hypothermia during caesarean section and postoperative infection

ELIGIBILITY:
Inclusion Criteria: Caesarean section surgery -

Exclusion Criteria: Stillborn baby, baby admitted to neonatal intensive care,

-

Ages: 18 Years to 50 Years | Sex: Female
Age Groups: Adult
Study Population: Females giving birth through caesarean section
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2030-11-01 (Estimated); Study Completion 2030-11-01 (Estimated)

PRIMARY OUTCOMES:
Patient reported recovery after caesarean delivery and symptoms of post caesarean infection | Data collection 24 hours after surgery and 7 days after surgery and 30 days after surgery
  Data collection using questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Reine, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo university hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided